CLINICAL TRIAL: NCT00467415
Title: Multi-Center Project: Supported Speed Treadmill Training Exercise Program (SSTTEP) for Marginally Ambulatory Children With Cerebral Palsy
Brief Title: Supported Speed Treadmill Training Exercise Program (SSTTEP) for Marginally Ambulatory Children With Cerebral Palsy
Acronym: SSTTEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Shriners Hospital for Children, Shriners Hospital for Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHC_COSAB9147
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Last update posted 2009-06-29 (Estimated); Status verified 2008-08

CONDITIONS: Cerebral Palsy
Keywords: Walking; Treadmill; Partial Weightbearing
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Partial body weight support treadmill training — Treadmill ambulation for 12 weeks. First 2 weeks for 10 total dose hours within clinical setting, final 10 weeks with 30 min/5 times week.
Behavioral: Exercise — Functional Strengthening exercise program for 12 weeks. First 2 weeks for 10 total dose hours within clinical setting, final 10 weeks with 30 min/5 times week.

SUMMARY:
The investigators are studying the effects of a 12-week exercise program, consisting of either:

1. Walking on a treadmill with partial body weight
2. Functional exercise program

The investigators would like to know the effects these two exercise programs have on the quality of life, muscle strength and control, coordination, walking, and functional movement of children with cerebral palsy who are marginal ambulators. This is a randomized control trial with subjects randomly assigned to one of the 2 groups.Subjects in both groups will be seen twice a day for two weeks at our hospital for intervention and parent training, and then participate in a 10 week home-based program. During each subject's two-week clinic-based training, a parent or caregiver is trained in all home program exercises and/or equipment usage. This person must be able to safely perform the exercise program with the child. Each subject will also need to participate in three separate 5-hour long data collection sessions scheduled over the 4 month study period.

DETAILED DESCRIPTION:
This project proposes to answer the following questions: Is partial body weight supported treadmill gait training (PBWSTT) effective in improving ambulation abilities, neuromuscular impairments, functional mobility, disability, and quality of life in marginally ambulatory children with cerebral palsy.

Specific Aim 1: Assess the effect of a PBWSTT locomotor training intervention on quality of life, treatment expectations, self-efficacy, and activity and participation of children with CP with limited ambulation skills. We hypothesize that in comparison to a control group, after a 12 week locomotor intervention, children with CP (intervention group) with limited ambulation skills will demonstrate greater improvements in scores from common questionnaires compared to the control group.

Specific Aim 2: Assess the effect of a PBWSTT locomotor training intervention on gross motor skills; physical function; biomechanics and coordination dynamics of ambulation; and physical activity in ambulatory children with CP. We hypothesize that in comparison to a control group, after a 12 week PBWSTT locomotor training intervention children with CP with limited ambulation skills will demonstrate greater improvements in functional test scores compared to the control group.

Specific Aim 3: Assess the effect of a PBWSTT locomotor training intervention on measures of body structure and function including: spasticity; muscle strength; and joint-specific motor control. We hypothesize that in comparison to a control group, after a 12 week PBWSTT locomotor training intervention children with CP with limited ambulation skills will demonstrate greater improvements in: muscle strength, spasticity and joint specific motor control compared to the control group.

This is a single blinded, randomized, controlled pre-test/post-test study design. Sixty six ambulatory children between the ages of 6-12 years of age with cerebral palsy will undergo a 12-week training program. Thirty three of these children will undergo a Supported Speed Treadmill Training Exercise Program (SSTTEP), and the remaining 33 children will receive the same amount of conventional physical therapy in the form of a personalized home exercise program and serve as a control group. Three sets of measures will be obtained: A1) at baseline prior to intervention; A2) at the end of the 12-week intervention period; and A3) 4 weeks after the intervention has ended.

The two primary aims of our study are to assess the efficacy of SSTTEP in improving quality of life, functional ambulation, energy expenditure, gross motor skills, and muscle strength and tone; and to assess the efficacy of SSTTEP in improving the coordination of stepping and ambulation in children with CP.

The intervention group will undergo a program of 10 hours of intensive SSTTEP training over a 14 day period. After the initial training, the subjects will participate in a home program of 30 minutes/5 times per week for an additional 10 weeks.

The control group with undergo a personalized exercise program consisting of 10 hours of intensive training over a 14 day period. After the initial training, the subjects will participate in a home program of 30 minutes/5 times per week for an additional 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of spastic cerebral palsy;
2. Impaired ambulation abilities as evidenced by a decreased in gait velocity below 80% of age expected value or gross motor function classification scale (GMFCS) Level III or IV;
3. Able to ambulate independently for 8 steps with/without assistive devices to allow for adequate motion analysis data collection;
4. Body weight of less than 150 pounds;
5. Between the ages of 6 and 13 years;
6. Able to follow multiple step commands and to attend to tasks associated with data collection;
7. Willingness to travel to one of the three sites for data collection sessions, and 2 weeks of intensive intervention;
8. Willingness to commit to home program 30 minutes per session, 5 times week for 10 weeks, as well as adequate space and supervision for treadmill use at home;
9. No reported musculoskeletal, cardiovascular or pulmonary conditions that would limit participation in moderate exercise program;
10. Minimum of 12 months post surgery including soft tissue releases
11. Six months post-Botox injections, significant changes in Baclofen dosing, or casting procedures to the lower extremities;
12. Passive range of motion of lower extremity joints: < 30º contracture of hip in extension as measured by the Thomas Test; passive dorsiflexion range of motion to -15º with the knee extended, and knee extension range (90º/90º test) to 70º and <-20º knee extension.
13. At least 2 years post- dorsal rhizotomy.

Exclusion Criteria:

1. Children with "mixed" types of CP (i.e. athetosis) or other movement disorders (e.g. ataxia);
2. Children receiving intrathecal Baclofen (baclofen pump);

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Gait Spatio-Temporal Parameters | 6 months
Muscle Activation and Timing | 6 months
Pediatric Quality of Life Inventory (PEDS-QL) | 6 months
Canadian Occupational Performance Measure (COPM) | 6 months
Children's Assessment of Participation and Enjoyment (CAPE) | 6 months
Piers-Harris Children's Self-Concept Scale, 2nd Edition (PHCSCS-2) | 6 months
Gross Motor Function Measure (GMFM) | 6 months
Pediatric Outcomes Data Collection Instrument (PODCI) | 6 months
Gait Velocity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Randal Betz, MD, Principal Investigator — Shriners Hospital for Children, Philadelphia
Locations (3):
- United States (3):
  - Shriners Hospital for Children, Shreveport, Shreveport, Louisiana
  - Washington University, St Louis, Missouri
  - Shriners Hospital for Children, Philadelphia, Philadelphia, Pennsylvania